CLINICAL TRIAL: NCT06677138
Title: A Phase 1 Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of Gefurulimab (ALXN1720) in Healthy Chinese Adults
Brief Title: PK Study of Gefurulimab SC in Healthy Chinese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6780C00003
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Chinese; gefurulimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gefurulimab (Experimental): Participants will receive a single SC dose of gefurulimab in the abdomen on Day 1.
  Interventions: Drug: gefurulimab

INTERVENTIONS:
Drug: gefurulimab — Participants will receive gefurulimab subcutaneously (SC).

SUMMARY:
The primary objective of this study is to characterize the PK properties of a single dose of gefurulimab in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 45 years of age, inclusive, at the time of signing the informed consent.
* Body weight within ≥ 45 kg to < 110 kg and BMI within the range 18 to 30 kg/m2 (inclusive) at Screening and Admission (Day -1).
* Participants who are healthy as determined by medical evaluation with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation.
* QTcF ≤ 450 msec for male participants and ≤ 460 msec for female participants at Screening and prior to dosing on Day 1.
* Documented vaccination against N meningitidis serotypes A, C, W-135, Y at least 28 days and not more than 3 years prior to dosing on Day 1.

Exclusion Criteria:

* History of any Neisseria meningitidis infection.
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders.
* Abnormal blood pressure as determined by the Investigator.
* History of latent or active TB (Tuberculosis) or exposure to endemic areas.
* Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing.
* History of latent or active TB or exposure to endemic areas within 8 weeks prior to the Screening Visit confirmed by QuantiFERON®-TB test.
* Significant allergies to humanized biologics.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions.
* History of clinically significant allergic reaction (eg, anaphylaxis or angioedema) to any product (eg, food, pharmaceutical).
* History of allergy or intolerance to penicillin or cephalosporin.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Current or chronic history of liver disease.
* Evidence of human immunodeficiency virus (HIV) infection (positive HIV type 1 or type 2 antibody).
* Evidence of hepatitis B infection (positive hepatitis B surface antigen [HBsAg] or positive total hepatitis B core antibody [HBcAb] with negative surface antibody [anti-HBs]), or hepatitis C viral infection (positive HCV RNA).
* Female participants who have a positive pregnancy test at Screening or Admission.
* Positive prestudy drug/alcohol screen; positive result may be repeated once.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of Gefurulimab | Day 1 predose through Day 92 postdose
Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Gefurulimab | Day 1 predose through Day 92 postdose

SECONDARY OUTCOMES:
Serum Free Complement Component 5 (C5) Concentration | Day 1 predose through Day 92 postdose
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day 1 through Day 92
Number of Participants With Anti-drug Antibodies (ADAs) | Day 1 through Day 92
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Associated With Prefilled Syringe With Needle Safety Device (PFS-SD) | Day 1 through Day 92
Number of Participants With Successful and Failed Dose Administrations | Day 1 through Day 92

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR